CLINICAL TRIAL: NCT03063086
Title: A Randomized, Double-blind, Double-dummy, Active-controlled, 3-period Complete Cross-over Study to Assess the Bronchodilator Effect and Safety of Two Doses of QVM149 Compared to a Fixed Dose Combination of Salmeterol/Fluticasone in Patients With Asthma
Brief Title: Assess Bronchodilator Effect and Safety of Two Doses of QVM149 Compared to a Fixed Dose Combination of Salmeterol/Fluticasone in Patients With Asthma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CQVM149B2208
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Results first posted 2019-12-13 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Active Comparator): A-B-C
  Interventions: Drug: QVM149 150/50/80 μg o.d.; Drug: QVM149 150/50/160 μg o.d.; Drug: salmeterol/fluticasone FDC 50/500 μg b.i.d.
- Sequence 2 (Active Comparator): A-C-B
  Interventions: Drug: QVM149 150/50/80 μg o.d.; Drug: QVM149 150/50/160 μg o.d.; Drug: salmeterol/fluticasone FDC 50/500 μg b.i.d.
- Sequence 3 (Active Comparator): B-C-A
  Interventions: Drug: QVM149 150/50/80 μg o.d.; Drug: QVM149 150/50/160 μg o.d.; Drug: salmeterol/fluticasone FDC 50/500 μg b.i.d.
- Sequence 4 (Active Comparator): B-A-C
  Interventions: Drug: QVM149 150/50/80 μg o.d.; Drug: QVM149 150/50/160 μg o.d.; Drug: salmeterol/fluticasone FDC 50/500 μg b.i.d.
- Sequence 5 (Active Comparator): C-A-B
  Interventions: Drug: QVM149 150/50/80 μg o.d.; Drug: QVM149 150/50/160 μg o.d.; Drug: salmeterol/fluticasone FDC 50/500 μg b.i.d.
- Sequence 6 (Active Comparator): C-B-A
  Interventions: Drug: QVM149 150/50/80 μg o.d.; Drug: QVM149 150/50/160 μg o.d.; Drug: salmeterol/fluticasone FDC 50/500 μg b.i.d.

INTERVENTIONS:
Drug: QVM149 150/50/80 μg o.d. — A
Drug: QVM149 150/50/160 μg o.d. — B
Drug: salmeterol/fluticasone FDC 50/500 μg b.i.d. — C

SUMMARY:
The purpose of this study is to assess peak FEV1 of two doses of QVM149 compared to a fixed-dose combination of salmeterol/fluticasone (50/500μg b.i.d.) and to characterize the respective 24 hour bronchodilator effect profiles in patients with asthma. Data from this study will complement lung function data obtained in the pivotal QVM149 phase 3 program by assessing the bronchodilatory effect of QVM149 at multiple time-points over an entire dosing interval of 24 hours.

ELIGIBILITY:
Key Inclusion criteria

* Male and female adult patients ≥ 18 years old and ≤ 75 years.
* Patients with a documented physician diagnosis of asthma for a period of at least 12 months prior to Visit 1 (Screening).
* Patients who have used ICS and LABA combinations for asthma for at least 3 month and at a stable medium or high dose of ICS for at least 1 month prior to Visit 1 (Screening).
* Pre-bronchodilator FEV1 of < 80 % of the predicted normal value at screening Visit 1 (spirometry will not be repeated at baseline prior to randomization).
* Patients who demonstrate an increase in FEV1 of ≥ 12 % and 200 mL after administration of 400 µg salbutamol/360 µg albuterol (or equivalent do se) at Visit 1 (Screening). All patients must perform a reversibility test at Visit 1 (Screening). If reversibility is not demonstrated at Visit 1 (Screening), then, reversibility testing may be repeated once during the screening period.
* If reversibility is not demonstrated at Visit 1 (retesting allowed once), patients must be screen failed. Spacer devices are not permitted during reversibility testing Key Exclusion criteria
* Patients who have smoked or inhaled tobacco products within the 6 month period prior to Visit 1
* Patients who have had an asthma attack/exacerbation requiring systemic steroids or hospitalization or emergency room visit within 6 weeks of Visit 1
* Patients with narrow-angle glaucoma, symptomatic benign prostatic hyperplasia (BPH) or bladder-neck obstruction or severe renal impairment or urinary retention
* Patients who have had a respiratory tract infection or asthma worsening within 4 weeks prior to Visit 1
* Patients with any chronic conditions affecting the upper respiratory tract
* Patients with a history of chronic lung diseases other than asthma, including (but not limited to) COPD, sarcoidosis, interstitial lung disease, cystic fibrosis, clinically significant bronchiectasis and active tuberculosis.
* Patients with Type I diabetes or uncontrolled Type II diabetes (HbA1c >9% at screening).
* Patients who have a clinically significant ECG abnormality at Visit 1
* Patients with a history of hypersensitivity or intolerance to any of the study drugs (including excipients)
* Patients with narcolepsy and/or insomnia.
* Patients on Maintenance Immunotherapy (desensitization) for allergies for less than 3 months prior to Visit 2 or patients on Maintenance Immunotherapy for more than 3 months prior to Visit 2 but expected to change throughout the course of the study.
* Pregnant or nursing (lactating) women
* Women of child-bearing potential must use Highly effective contraception methods
* Patients who have discontinued LAMA therapy in the past for any safety, tolerability or perceived lack of efficacy reason.
* History of paradoxical bronchospasm in response to inhaled medicines.
* Patients with a history of clinically relevant bronchoconstriction upon repeated forced expiratory maneuvers.
* Patient with a serum potassium level below the laboratory limit of normal at screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-01-21 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- Novartis Investigative Site, Sofia, Bulgaria
- China (3):
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Shanghai
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Wiesbaden
- Novartis Investigative Site, Groningen, GZ, Netherlands
- Novartis Investigative Site, Bucharest, Romania
- Novartis Investigative Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=392

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1 (A-B-C): QVM149 150/50/80 μg o.d; QVM149 150/50/160 μg o.d; salmeterol/fluticasone FDC 50/500 μg b.i.d.
- Sequence 2(A-C-B): QVM149 150/50/80 μg o.d; salmeterol/fluticasone FDC 50/500 μg b.i.d.; QVM149 150/50/160 μg o.d;
- Sequence 3(B-C-A): QVM149 150/50/160 μg o.d; salmeterol/fluticasone FDC 50/500 μg b.i.d.; QVM149 150/50/80 μg o.d
- Sequence 4(B-A-C): QVM149 150/50/160 μg o.d; QVM149 150/50/80 μg o.d; salmeterol/fluticasone FDC 50/500 μg b.i.d
- Sequence 5(C-A-B): salmeterol/fluticasone FDC 50/500 μg b.i.d; QVM149 150/50/80 μg o.d; QVM149 150/50/160 μg o.d
- Sequence 6(C-B-A): salmeterol/fluticasone FDC 50/500 μg b.i.d.; QVM149 150/50/160 μg o.d; QVM149 150/50/80 μg o.d
Period: Overall Study
Arm/Group | Sequence 1 (A-B-C) | Sequence 2(A-C-B) | Sequence 3(B-C-A) | Sequence 4(B-A-C) | Sequence 5(C-A-B) | Sequence 6(C-B-A)
Started | 19 | 20 | 18 | 20 | 20 | 19
Completed | 16 | 19 | 17 | 17 | 20 | 18
Not Completed | 3 | 1 | 1 | 3 | 0 | 1
Not completed — technical problems | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 1 | 1 | 0 | 0
Not completed — subject/guardian decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance with study treatment | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants randomized to one of six treatment sequences
Arm/Group | All Participants
Number analyzed (Participants) | 116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.5 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 106
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Peak FEV1 (L) Defined as the Highest Bronchodilatory Effect on FEV1 During a Period of 5 Min to 4 h After the Last Evening Dose of Each Treatment Period
Description: The highest bronchodilator effect on FEV1 during a period of 5 min to 4 h after the last evening dose of each treatment period . To demonstrate superiority in peak bronchodilator effect of QVM149 at a dose of 150/50/160 μg o.d. and 150/50/80 μg o.d. compared to a FDC of salmeterol/fluticasone at a dose of 50/500 μg b.i.d. after 3 weeks of treatment in patients with asthma
Time Frame: 3 weeks
Population: Pharmacodynamics set - The PD analysis set included all patients with any available PD data, who received any study treatment and experienced no protocol deviations with relevant impact on PD data.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- QVM149 150/50/160 μg o.d.: QVM149 150/50/160 μg o.d.
- QVM149 150/50/80 μg o.d.: QVM149 150/50/80 μg o.d.
- Salmeterol/Fluticasone 50/500 µg b.i.d: salmeterol/fluticasone 50/500 µg b.i.d
Arm/Group | QVM149 150/50/160 μg o.d. | QVM149 150/50/80 μg o.d. | Salmeterol/Fluticasone 50/500 µg b.i.d
Number analyzed (Participants) | 112 | 115 | 111
Liters | 2.792 (0.0750) | 2.779 (0.0750) | 2.620 (0.0750)
Statistical Analysis 1: Comparison: QVM149 150/50/160 μg o.d; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.172, 95% CI 2-sided [0.137 to 0.208]
Statistical Analysis 2: Comparison: QVM149 150/50/80 μg o.d; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Median Difference (Final Values) = 0.159, 95% CI 2-sided [0.123 to 0.195]

2. Secondary Outcome: FEV1 Over 24 h After 21 Days of Treatment in Relation to Evening Dose
Description: To evaluate the bronchodilator effect of each dose of QVM149 compared to salmeterol/fluticasone FDC after 3 weeks of treatment at -45 min, -15 min, 5 min, 15 min, 30 min, 1 h, 2 h, 3h, 4 h, 8 h, 10 h, 11 h 55 min, 14 h, 18 h, 21 h, 23 h 15 min, 23 h 45 min.
Time Frame: -45 min, -15 min, 5 min, 15 min, 30 min, 1 h, 2 h, 3h, 4 h, 8 h, 10 h, 11 h 55 min, 14 h, 18 h, 21 h, 23 h 15 min, 23 h 45 min at 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVM149 150/50/160 μg o.d. | QVM149 150/50/80 μg o.d. | Salmeterol/Fluticasone 50/500 µg b.i.d
Number analyzed (Participants) | 112 | 115 | 111
Liters
  -45 min: number analyzed (Participants) | 111 | 111 | 111
  -45 min | 2.6237 (0.07505) | 2.5639 (0.07503) | 2.4931 (0.07505)
  -15 min: number analyzed (Participants) | 111 | 109 | 109
  -15 min | 2.6023 (0.07479) | 2.5630 (0.07478) | 2.4835 (0.07480)
  5 min: number analyzed (Participants) | 110 | 108 | 109
  5 min | 2.6412 (0.07446) | 2.6179 (0.07445) | 2.5035 (0.07446)
  15 min: number analyzed (Participants) | 110 | 108 | 108
  15 min | 2.6696 (0.07531) | 2.6137 (0.07532) | 2.5172 (0.07533)
  30 min: number analyzed (Participants) | 110 | 108 | 110
  30 min | 2.6873 (0.07444) | 2.6504 (0.07444) | 2.5286 (0.07444)
  1 h: number analyzed (Participants) | 110 | 107 | 108
  1 h | 2.6922 (0.07430) | 2.6825 (0.07431) | 2.5398 (0.07431)
  2 h: number analyzed (Participants) | 109 | 107 | 107
  2 h | 2.7033 (0.07441) | 2.6996 (0.07443) | 2.5244 (0.07443)
  3 h: number analyzed (Participants) | 109 | 107 | 106
  3 h | 2.6995 (0.07449) | 2.6719 (0.07450) | 2.5296 (0.07451)
  4 h: number analyzed (Participants) | 109 | 107 | 106
  4 h | 2.6815 (0.07482) | 2.6565 (0.07484) | 2.5164 (0.07485)
  8 h: number analyzed (Participants) | 109 | 104 | 105
  8 h | 2.6801 (0.07454) | 2.6550 (0.07459) | 2.4918 (0.07459)
  10 h: number analyzed (Participants) | 108 | 105 | 105
  10 h | 2.6999 (0.07489) | 2.6796 (0.07494) | 2.4908 (0.07495)
  11h 55 min: number analyzed (Participants) | 107 | 104 | 103
  11h 55 min | 2.7042 (0.07486) | 2.6641 (0.07490) | 2.4841 (0.07491)
  14 h: number analyzed (Participants) | 107 | 103 | 103
  14 h | 2.6829 (0.07456) | 2.6541 (0.07459) | 2.5354 (0.07461)
  18 h: number analyzed (Participants) | 107 | 102 | 102
  18 h | 2.6345 (0.07451) | 2.6073 (0.07455) | 2.5329 (0.07457)
  21 h: number analyzed (Participants) | 107 | 102 | 100
  21 h | 2.6113 (0.07466) | 2.5989 (0.07472) | 2.5133 (0.07475)
  23 h 15 min: number analyzed (Participants) | 105 | 100 | 100
  23 h 15 min | 2.6143 (0.07433) | 2.5950 (0.07438) | 2.4854 (0.07439)
  23 h 45 min: number analyzed (Participants) | 105 | 99 | 100
  23 h 45 min | 2.5966 (0.07433) | 2.5722 (0.07438) | 2.4913 (0.07439)

3. Secondary Outcome: FVC Over 24 h After 21 Days of Treatment in Relation to Evening Dose
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- Salmeterol/Fluticasone 50/500 μg b.i.d: Salmeterol/fluticasone 50/500 μg b.i.d
Arm/Group | QVM149 150/50/160 μg o.d. | QVM149 150/50/80 μg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d
Number analyzed (Participants) | 112 | 115 | 111
Liters
  -45min: number analyzed (Participants) | 111 | 110 | 110
  -45min | 3.9046 (1.03169) | 3.8538 (0.98086) | 3.7626 (1.00067)
  -15min: number analyzed (Participants) | 111 | 109 | 108
  -15min | 3.8743 (1.04318) | 3.8571 (0.97420) | 3.7230 (0.94180)
  5min: number analyzed (Participants) | 110 | 107 | 107
  5min | 3.8656 (0.99877) | 3.8976 (1.00323) | 3.7536 (0.93696)
  15min: number analyzed (Participants) | 110 | 107 | 106
  15min | 3.8669 (0.98489) | 3.8971 (0.96840) | 3.7290 (0.94033)
  30min: number analyzed (Participants) | 109 | 108 | 108
  30min | 3.8700 (0.99289) | 3.9002 (0.99091) | 3.7695 (0.96026)
  1h: number analyzed (Participants) | 109 | 107 | 107
  1h | 3.8756 (0.99978) | 3.8993 (0.99141) | 3.7530 (0.97083)
  2h: number analyzed (Participants) | 108 | 107 | 107
  2h | 3.8698 (0.99623) | 3.8985 (0.99369) | 3.7629 (0.97164)
  3h: number analyzed (Participants) | 109 | 106 | 105
  3h | 3.8576 (0.98598) | 3.8766 (0.97806) | 3.7575 (0.96899)
  4h: number analyzed (Participants) | 109 | 107 | 106
  4h | 3.8744 (0.99833) | 3.8627 (0.95673) | 3.7629 (0.98205)
  8h: number analyzed (Participants) | 109 | 103 | 105
  8h | 3.9020 (0.98241) | 3.9217 (0.99184) | 3.7683 (1.00410)
  10h: number analyzed (Participants) | 108 | 103 | 105
  10h | 3.8976 (0.98360) | 3.9504 (0.99286) | 3.7809 (0.98213)
  11h 55min: number analyzed (Participants) | 107 | 102 | 102
  11h 55min | 3.9271 (0.98924) | 3.9405 (1.00198) | 3.7911 (0.99102)
  14h: number analyzed (Participants) | 107 | 103 | 103
  14h | 3.9091 (1.00241) | 3.9210 (0.97942) | 3.8089 (1.02918)
  18h: number analyzed (Participants) | 107 | 102 | 101
  18h | 3.8675 (0.95725) | 3.9151 (1.02198) | 3.7824 (0.98395)
  21h: number analyzed (Participants) | 107 | 101 | 100
  21h | 3.8438 (1.00672) | 3.8694 (0.98786) | 3.7680 (1.00768)
  23h 15min: number analyzed (Participants) | 104 | 100 | 100
  23h 15min | 3.7997 (0.97550) | 3.8673 (0.99915) | 3.7395 (1.01764)
  23h 45min: number analyzed (Participants) | 105 | 99 | 98
  23h 45min | 3.8034 (0.99036) | 3.8603 (0.98502) | 3.7431 (1.00668)

4. Secondary Outcome: FEV1/FVC Ratio Over 24 h After 21 Days of Treatment in Relation to Evening Dose
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | QVM149 150/50/160 μg o.d. | QVM149 150/50/80 μg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d
Number analyzed (Participants) | 112 | 115 | 111
Ratio
  -45min: number analyzed (Participants) | 107 | 107 | 108
  -45min | 0.6701 (0.10880) | 0.6612 (0.10358) | 0.6527 (0.10867)
  -15min: number analyzed (Participants) | 107 | 106 | 108
  -15min | 0.6707 (0.10646) | 0.6669 (0.10422) | 0.6539 (0.10526)
  5min: number analyzed (Participants) | 109 | 106 | 103
  5min | 0.6788 (0.10300) | 0.6754 (0.10370) | 0.6563 (0.10639)
  15min: number analyzed (Participants) | 106 | 103 | 103
  15min | 0.6873 (0.10126) | 0.6778 (0.10734) | 0.6560 (0.10823)
  30min: number analyzed (Participants) | 106 | 103 | 108
  30min | 0.6878 (0.10137) | 0.6844 (0.10699) | 0.6573 (0.10552)
  1h: number analyzed (Participants) | 108 | 106 | 105
  1h | 0.6900 (0.09764) | 0.6895 (0.09940) | 0.6632 (0.10403)
  2h: number analyzed (Participants) | 107 | 105 | 106
  2h | 0.6939 (0.09629) | 0.6932 (0.10073) | 0.6647 (0.10413)
  3h: number analyzed (Participants) | 108 | 106 | 104
  3h | 0.6968 (0.10159) | 0.6890 (0.10052) | 0.6634 (0.10436)
  4h: number analyzed (Participants) | 106 | 107 | 105
  4h | 0.6897 (0.10060) | 0.6879 (0.09733) | 0.6605 (0.10419)
  8h: number analyzed (Participants) | 105 | 95 | 102
  8h | 0.6842 (0.10782) | 0.6802 (0.11349) | 0.6492 (0.10814)
  10h: number analyzed (Participants) | 105 | 99 | 104
  10h | 0.6916 (0.10550) | 0.6858 (0.10468) | 0.6489 (0.11155)
  11h 55min: number analyzed (Participants) | 103 | 99 | 102
  11h 55min | 0.6853 (0.10672) | 0.6791 (0.10656) | 0.6482 (0.10810)
  14h: number analyzed (Participants) | 104 | 101 | 101
  14h | 0.6846 (0.10842) | 0.6848 (0.10450) | 0.6567 (0.11048)
  18h: number analyzed (Participants) | 104 | 101 | 97
  18h | 0.6801 (0.09943) | 0.6741 (0.10240) | 0.6546 (0.10369)
  21h: number analyzed (Participants) | 106 | 99 | 99
  21h | 0.6790 (0.10890) | 0.6785 (0.10387) | 0.6562 (0.10729)
  23h 15min: number analyzed (Participants) | 102 | 98 | 100
  23h 15min | 06821 (0.10386) | 0.6791 (0.09986) | 0.6548 (0.10423)
  23h 45min: number analyzed (Participants) | 104 | 98 | 98
  23h 45min | 0.6782 (0.10457) | 0.6776 (0.10111) | 0.6537 (0.10934)

5. Secondary Outcome: FEV1 AUC 5 Min - 1 h (Day 21) FEV1 AUC 5 Min - 4 h (Day 21) and FEV1 AUC 5 Min - 23 h 45 Min (Day 21)
Description: To evaluate the bronchodilator effect of each dose of QVM149 compared to salmeterol/ fluticasone FDC by measuring standardized FEV1 AUCs after 3 weeks of treatment respective period.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVM149 150/50/160 μg o.d. | QVM149 150/50/80 μg o.d. | Salmeterol/Fluticasone 50/500 µg b.i.d
Number analyzed (Participants) | 112 | 115 | 111
Liters
  FEV1 AUC 5 min - 1 h: number analyzed (Participants) | 108 | 103 | 100
  FEV1 AUC 5 min - 1 h | 2.673 (0.0735) | 2.644 (0.0736) | 2.513 (0.0737)
  FEV1 AUC 5 min - 4 h: number analyzed (Participants) | 104 | 104 | 99
  FEV1 AUC 5 min - 4 h | 2.687 (0.0741) | 2.669 (0.0741) | 2.510 (0.0742)
  FEV1 AUC 5 min - 23 h 45 min: number analyzed (Participants) | 101 | 93 | 92
  FEV1 AUC 5 min - 23 h 45 min | 2.677 (0.0766) | 2.652 (0.0768) | 2.515 (0.0768)

6. Secondary Outcome: Trough FEV1 After 21 Days of Treatment
Description: To evaluate post-dose trough bronchodilator effect of each dose of QVM149 compared to salmeterol/fluticasone FDC after 3 weeks of treatment in the respective treatment period. The trough FEV1 is the mean value of FEV1 at 23 h 15 min and 23 h 45 min post-dose
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVM149 150/50/160 μg o.d. | QVM149 150/50/80 μg o.d. | Salmeterol/Fluticasone 50/500 µg b.i.d
Number analyzed (Participants) | 112 | 115 | 111
Liters | 2.623 (0.0756) | 2.6046 (0.0757) | 2.4998 (0.0757)
Statistical Analysis 1: Comparison: QVM149 150/50/160 μg o.d; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.124, 95% CI 2-sided [0.086 to 0.161]

ADVERSE EVENTS:
Time Frame: Up to 22 days
Groups:
- QVM149 150/50/160 µg o.d.: QVM149 150/50/160 µg o.d.
- QVM149 150/50/80 µg o.d.: QVM149 150/50/80 µg o.d.
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | Salmeterol/Fluticasone 50/500 µg b.i.d.
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/115 | 0/111
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/115 | 0/111
Other Adverse Events (participants affected / at risk) | 14/112 | 18/115 | 21/111
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVM149 150/50/160 µg o.d. (N=112) | QVM149 150/50/80 µg o.d. (N=115) | Salmeterol/Fluticasone 50/500 µg b.i.d. (N=111)
Nasopharyngitis (Infections and infestations) | 3 | 7 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 10 | 10 | 13
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Study Protocol (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT03063086/Prot_001.pdf
  • Statistical Analysis Plan (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT03063086/SAP_000.pdf